CLINICAL TRIAL: NCT01141439
Title: A Retrospective Evaluation of the Effectiveness and Cost-effectiveness of HFA-BDP MDI (Qvar®) Compared With CFC-BDP MDI and FP MDI Used in the Management of Asthma in a Representative UK UK Primary Care Population
Brief Title: Real-world Effectiveness and Cost-effectiveness of Leading Inhaled Corticosteroids in Asthma Management
Acronym: QvarAsthma
Status: Completed | Type: Observational
Sponsor: Research in Real-Life Ltd (Network)
Collaborators: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Professor David Price, Research in Real Life Limited
Other Study IDs: BA4
Record Dates: First submitted 2010-06-09; First posted 2010-06-10 (Estimated); Last update posted 2013-03-14 (Estimated); Status verified 2013-03

CONDITIONS: Asthma
Keywords: Primary care; Asthma management; Inhaled corticosteroids; Beclomethasone dipropionate; Fluticasone propionate; Metred dose inhaler; Extra-fine hydrofluoroalkane; Chlorofluorocarbon
MeSH Terms: conditions — Asthma | interventions — Beclomethasone; Fluticasone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (6):
- IPDI HFA-BDP MDI: Patients who commenced inhaled corticosteroid therapy as HFA-BDP via MDI
  Interventions: Drug: Extra-fine hydrofluoroalkane-beclomethasone dipropionate
- IPDI FP MDI: Patients who commenced inhaled corticosteroid therapy as FP via MDI
  Interventions: Drug: fluticasone propionate
- IPDA FP MDI: Patients who had a step up in inhaled corticosteroid therapy as FP via MDI
  Interventions: Drug: Fluticasone propionate
- IPDA HFA-BDP MDI: Patients who had a step up in inhaled corticosteroid therapy as HFA-BDP via MDI
  Interventions: Drug: Extra-fine hydrofluoroalkane-beclomethasone dipropionate
- IPDI CFC-BDP MDI: Patients who commenced inhaled corticosteroid therapy as CFC-BDP via MDI
  Interventions: Drug: Chlorofluorocarbon beclomethasone dipropionate
- IPDA CFC-BDP MDI: Patients who had a step up in inhaled corticosteroid therapy as CFC-BDP via MDI
  Interventions: Drug: Beclomethasone dipropionate

INTERVENTIONS:
Drug: Extra-fine hydrofluoroalkane-beclomethasone dipropionate — Initiation of HFA-BDP (any dose) in steroid naive patients via MDI
  Other Names: Qvar®
  Groups: IPDI HFA-BDP MDI
Drug: Extra-fine hydrofluoroalkane-beclomethasone dipropionate — An increase in the baseline BDP-equivalent dose of inhaled corticosteroid as HFA-BDP via MDI
  Other Names: Qvar
  Groups: IPDA HFA-BDP MDI
Drug: Fluticasone propionate — An increase in the baseline BDP-equivalent dose of inhaled corticosteroid as FP via MDI
  Groups: IPDA FP MDI
Drug: Beclomethasone dipropionate — An increase in the baseline BDP-equivalent dose of inhaled corticosteroid as CFC-BDP via MDI
  Groups: IPDA CFC-BDP MDI
Drug: fluticasone propionate — Initiation of FP (any dose) via MDI in steroid naive patient
  Groups: IPDI FP MDI
Drug: Chlorofluorocarbon beclomethasone dipropionate — Initiation of CFC-BDP (any dose) via MDI in steroid naive patient
  Groups: IPDI CFC-BDP MDI

SUMMARY:
The objective of the study was to compare the effectiveness, cost-effectiveness and direct healthcare costs of managing asthma in patients with evidence of persistent asthma, following the initiation and increased dose of inhaled corticosteroid (ICS) therapy using HFA-BDP (Qvar®) (either as initial therapy or as a step-up therapy) compared with the most commonly prescribed alternative ICS in the UK, CFC-beclometasone (BDP) and fluticasone (FP) as metered dose inhalers (MDIs). Qvar vs FP analyses were split between adults (12-60yrs) and paediatrics (5-11yrs).

DETAILED DESCRIPTION:
While current UK asthma guidelines are underpinned with evidence from RCTs, much of this evidence has been undertaken in patients who are not representative of the majority of the current UK asthma population. In fact it has been estimated that fewer than 10% of the patients seen in everyday clinical practice would be eligible for inclusion in such trials. The poor representation of the asthma population is due to a number of factors, such as tightly-controlled inclusion criteria for RCTs. There is therefore a need for more representative RCTs and real-life and observational studies to inform existing guidelines and help optimise asthma outcomes. A more holistic approach to respiratory research would see RCT evidence complimented by "real-life" data from pragmatic trials and observational studies.

A number of trends are emerged in asthma prescribing that warrant further investigation to ascertain their benefit to both the patient and the NHS. In particular, significant pressure exists to use the cheapest inhaler devices and formulations. An analysis of a pragmatic trial of Qvar versus standard CFC-BDP undertaken by Research in Real Life suggested that Qvar may be offer greater effectiveness in.5,6 In light of these data, the following report details the findings of a study designed to examine the effectiveness of Qvar in real-life clinical practice using the General Practice Research Database (GPRD).

ELIGIBILITY:
Inclusion Criteria:

Included patients must:

* aged 5-60 years
* evidence of asthma: a diagnostic code of asthma or ≥2 prescriptions for asthma in baseline year at different points in time including one of ICS
* on current therapy at the IPD, defined as ≥1 ICS script and ≥1 other asthma prescriptions in the 12 months prior to first change in therapy
* had definite dosing instructions
* have at least 1 year of up-to-standard (UTS) baseline data before IPD
* have at least 1 year of UTS outcome data after IPD.

Exclusion Criteria:

* had a diagnostic read code for chronic obstructive pulmonary disease (COPD) at any time
* had a diagnostic read code for chronic respiratory disease at any time
* For the therapy increase patient cohort, any patients receiving a combination inhaler in addition to their separate ICS inhaler in the year prior to IPD were also excluded.

Ages: 5 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Primary care asthma patients receiving who either initiated ICS therapy as any of extrafine HFA-BDP, CFC-BDP of FP via MDI at an index prescription date (IPD), or were on existing ICs therapy (any) and had an increase in ICS dose at IPD as any of extrafine HFA-BDP, CFC-BDP of FP via MDI
Sampling Method: Non-Probability Sample
Enrollment: 815377 (Actual)
Dates: Start 2001-01; Primary Completion 2007-06 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Proxy asthma control | One-year outcome period
  Primary composite measure asthma control defined as:
  * No recorded hospital attendance for asthma including admission, Accident & Emergency (A&E) attendance, out of hours attendance or Out-Patient Department (OPD) attendance, AND
  * No prescriptions for oral steroid, AND
  * No consultations, hospital admissions or A&E attendance for lower respiratory tract infections (LRTI) requiring antibiotics.

SECONDARY OUTCOMES:
Revised asthma control | One-year outcome period
  A revised definition of proxy asthma control for sensitivity analysis was defined as:
  * No recorded hospital attendance for asthma including admission, A&E attendance, out of hours attendance or OPD attendance, AND
  * No prescriptions for oral steroid, AND
  * No consultations, hospital admissions or A&E attendance for lower respiratory tract infections (LRTI) requiring antibiotics
  * Average daily prescribed dose of salbutamol of no more than 200mcg and terbutaline 500mcg.
Disaggregated components of the primary control outcome | One-year outcome period
  * Hospital admissions for asthma
  * Consultations and hospital attendances for LRTI requiring antibiotics
  * Prescriptions for oral steroids
  * SABA use
Time to the first asthma exacerbation | One-year outcome period
  Where an exacerbation is defined as:
  * An occurrence of unscheduled hospital admission/A&E attendances for asthma AND/OR
  * Use of oral steroids.
Success of the therapeutic regimen | One-year outcome period
  Defined as:
  * Exacerbation AND/OR
  * Increase in dose of ICS AND/OR
  * Change in ICS drug type AND/OR
  * Change in delivery device AND/OR
  * Use of additional therapy as defined by: LABAs, oral steroids, theophylline, leukotriene receptor antagonists (LTRAs)
Use of anti-fungals | One-year
  defined as incidences of definite oral candidiasis
Daily dose of ICS (BDP equivalent) at week 52 compared with week 0 and proportion on original dose of BDP Daily dose* of ICS (BDP equivalent) at week 52 compared with week 0 and proportion on original dose of BDP. | One-year outcome period
  BDP-equivalent dose were calculated by multiplying the Qvar and FP doses by a factor of 2. The dose at week 52 was compared with that at week 0 in order to identify the proportion of original (week 0) ICS dose.

CONTACTS AND LOCATIONS:
Overall Officials: David Price, Prof. MD, Principal Investigator — Company Director; Alison Chisholm, MSc, Study Director — Research Project Director
Locations (1):
- General Practice Research Database, London, London, United Kingdom

REFERENCES:
- [Background] Herland K, Akselsen JP, Skjonsberg OH, Bjermer L. How representative are clinical study patients with asthma or COPD for a larger "real life" population of patients with obstructive lung disease? Respir Med. 2005 Jan;99(1):11-9. doi: 10.1016/j.rmed.2004.03.026. PMID 15672843
- [Background] Travers J, Marsh S, Caldwell B, Williams M, Aldington S, Weatherall M, Shirtcliffe P, Beasley R. External validity of randomized controlled trials in COPD. Respir Med. 2007 Jun;101(6):1313-20. doi: 10.1016/j.rmed.2006.10.011. Epub 2006 Nov 17. PMID 17113277
- [Background] Thomas M, Cleland J, Price D. Database studies in asthma pharmacoeconomics: uses, limitations and quality markers. Expert Opin Pharmacother. 2003 Mar;4(3):351-8. doi: 10.1517/14656566.4.3.351. PMID 12614187
- [Background] Tannen RL, Weiner MG, Xie D. Use of primary care electronic medical record database in drug efficacy research on cardiovascular outcomes: comparison of database and randomised controlled trial findings. BMJ. 2009 Jan 27;338:b81. doi: 10.1136/bmj.b81. PMID 19174434
- [Background] Juniper EF, Price DB, Stampone PA, Creemers JP, Mol SJ, Fireman P. Clinically important improvements in asthma-specific quality of life, but no difference in conventional clinical indexes in patients changed from conventional beclomethasone dipropionate to approximately half the dose of extrafine beclomethasone dipropionate. Chest. 2002 Jun;121(6):1824-32. doi: 10.1378/chest.121.6.1824. PMID 12065345
- [Background] Price D, Haughney J, Duerden M, Nicholls C, Moseley C. The cost effectiveness of chlorofluorocarbon-free beclomethasone dipropionate in the treatment of chronic asthma: a cost model based on a 1-year pragmatic, randomised clinical study. Pharmacoeconomics. 2002;20(10):653-64. doi: 10.2165/00019053-200220100-00002. PMID 12162754
- [Background] Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis. 1987;40(5):373-83. doi: 10.1016/0021-9681(87)90171-8. PMID 3558716
- [Background] Cliniclue [homepage on the internet]. The Clinical Information Consultancy CLINICLUE® [updated 2008; cited 15 May 2009]. Available online at: http://www.cliniclue.com
- [Background] SPSS [homepage on the internet]. Chicago: SPSS Inc [updated 2009; cited 15 May 2009]. Available online at: http://www.spss.com/UK/
- [Background] Microsoft office online [homepage on the internet]. USA: Microsoft Corporation [updated 2009; cited 15 May 2009]. Available online at: http://office.microsoft.com/excel
- [Background] STATA: Data Analysis and Statistical Software [homepage on the internet]. Texas: STATA [updated 2009; cited 15 May 2009]. Available online at: http://www.stata.com/
- See also: Optimum Patient Care is the Research in Real Life's sister company (a social enterprise organisation) — http://www.optimumpatientcare.org